CLINICAL TRIAL: NCT05349136
Title: Effectiveness of Synchronous and Asynchronous Telerehabilitation-Based Action Observation Treatment in Children with Hemiparetic Cerebral Palsy
Brief Title: Telerehabilitation-Based Action Observation Treatment in Children with Hemiparetic Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Hilal Başak Can, Research Assistant, Marmara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09.2020.1353
Record Dates: First submitted 2022-04-05; First posted 2022-04-27 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2022-04

CONDITIONS: Hemiparetic Cerebral Palsy
Keywords: Cerebral Palsy; Hemiparesis; Telerehabilitation; Action Observation Treatment
MeSH Terms: conditions — Cerebral Palsy; Paresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Synchronous telerehabilitation group (Experimental): Synchronous telerehabilitation based-Action Observation Treatment and conventional physiotherapy
  Interventions: Other: Synchronous telerehabilitation group
- Asynchronous telerehabilitation group (Experimental): Asynchronous telerehabilitation based-Action Observation Treatment and conventional physiotherapy
  Interventions: Other: Asynchronous telerehabilitation group
- Control group (No Intervention): Conventional physiotherapy

INTERVENTIONS:
Other: Synchronous telerehabilitation group — This group will receive Action Observation Treatment with a synchronous telerehabilitation method. Children in this group will be applied Action Observation Treatment 5 days a week for 3 weeks, for a total of 15 sessions under the supervision of a physiotherapist via videoconferencing.
  Arms: Synchronous telerehabilitation group
Other: Asynchronous telerehabilitation group — This group will receive Action Observation Treatment with an asynchronous telerehabilitation method. Children in this group will be applied Action Observation Treatment 5 days a week for 3 weeks, for a total of 15 sessions under parental supervision.
  Arms: Asynchronous telerehabilitation group

SUMMARY:
The aim of this study is to evaluate the effectiveness of action observation therapy applied using two different telerehabilitation techniques (synchronous and asynchronous) to children with hemiparetic cerebral palsy.

DETAILED DESCRIPTION:
Action observation treatment (AOT) is a new rehabilitation technique. AOT involves the observation of purposeful actions, presented through a video-clip or performed by an operator, in order to imitate and then perform them. In this study, AOT will be applied by observing actions to be presented via video-clips. 36 children with hemiparetic cerebral palsy who meet the inclusion criteria and agree to participate in the study will be included. The participants will be randomly divided into three groups. The groups are: a) the synchronous telerehabilitation group, where AOT will be applied under the supervision of a physiotherapist via videoconferencing; b) the asynchronous telerehabilitation group, where AOT will be applied under parental supervision; and c) control group. Both the synchronous telerehabilitation group and the asynchronous telerehabilitation group will receive AOT 5 days a week for 3 weeks, for a total of 15 sessions, in addition to conventional physiotherapy. The control group will only receive conventional physiotherapy. A total of three evaluations will be made at baseline (T0), at the end of treatment (T1), and at two months of follow-up (T2).

ELIGIBILITY:
Inclusion Criteria:

* Presence of confirmed hemiparetic cerebral palsy
* Manual Ability Classification System ≤ 3
* Age between 6 and 12
* Absence of major visual and/or auditory deficits
* Sufficient cooperation to comprehend and complete the test procedure and participate in treatment
* House Functional Classification Score ≥4
* Grade ≤2 on the Modified Ashworth Scale

Exclusion Criteria:

* Seizures uncontrolled by therapy
* Surgery and/or botulinum toxin-A injections in the upper limb within 6 months prior to the baseline assessment
* Having a disabling behavioral disorder to treatment

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2022-11-09 (Actual); Primary Completion 2024-09-17 (Actual); Study Completion 2024-09-17 (Actual)

PRIMARY OUTCOMES:
Changes in Assisting Hand Assessment | Baseline (T0, 1 week before beginning of the study); T1 (within 1 week after the end of the treatment/control period); T2 (8 weeks after the end of the treatment/control period)
  The children's the assisting hand use in activities requiring bimanual use will be evaluated with the Assisting Hand Assessment. The game, which can be performed in a time frame of 10-15 minutes, will be recorded. Then the video will be watched. Twenty-two components regarding general use, arm use, grasp and release, fine motor adjustment, coordination, and pace of the performance will be scored on a four-point scale.

SECONDARY OUTCOMES:
Changes in Box and Blocks Test | Baseline (T0, 1 week before beginning of the study); T1 (within 1 week after the end of the treatment/control period); T2 (8 weeks after the end of the treatment/control period)
  The children's unilateral gross manual dexterity will be evaluated with the Box and Blocks Test, which is a timed test. First, the dominant hand will be asked to place the blocks from one side of the box to the other in 1 minute. The number of blocks placed on the other side of the box is recorded. Then it will be repeated with the other hand. The test can be completed in less than 10 minutes.
Changes in Minnesota Manual Dexterity Test | Baseline (T0, 1 week before beginning of the study); T1 (within 1 week after the end of the treatment/control period); T2 (8 weeks after the end of the treatment/control period)
  The children's manual dexterity required to turn and/or place disks with one or both hands will be assessed with the Minnesota Manual Dexterity Test. The completion time of the tasks will be recorded.
Changes in Children's Hand-use Experience Questionnaire | Baseline (T0, 1 week before beginning of the study); T1 (within 1 week after the end of the treatment/control period); T2 (8 weeks after the end of the treatment/control period)
  The children's use of assisting hands in various bimanual activities will be assessed with the Children's Hand-use Experience Questionnaire. This questionnaire will be completed by their parents.
Changes in ABILHAND-kids | Baseline (T0, 1 week before beginning of the study); T1 (within 1 week after the end of the treatment/control period); T2 (8 weeks after the end of the treatment/control period)
  The children's ease or difficulty in performing bimanual activities will be assessed with the ABILHAND-kids, which is a parent questionnaire.
Changes in Participation and Environment Measure - Children and Youth | Baseline (T0, 1 week before beginning of the study); T1 (within 1 week after the end of the treatment/control period); T2 (8 weeks after the end of the treatment/control period)
  The children's participation in the home, at school, and in the community will be assessed with the Participation and Environment Measure-Children and Youth, which is a parent questionnaire.
Changes in Trunk Impairment Scale | Baseline (T0, 1 week before beginning of the study); T1 (within 1 week after the end of the treatment/control period); T2 (8 weeks after the end of the treatment/control period)
  The children's static sitting balance, dynamic sitting balance, and trunk coordination will be assessed with the Trunk Impairment Scale. The total score is between 0-23. A higher score indicates better performance.
Treatment Satisfaction Assessed by the Visual Analog Scale | T1 (within 1 week after the end of the treatment/control period)
  The children and their parents' treatment satisfaction will be assessed separately with the visual analog scale. The value is between 0-10. A higher value indicates better satisfaction.
Treatment Satisfaction Assessed by the Visual Analog Scale | T2 (8 weeks after the end of the treatment/control period)
  The children and their parents' treatment satisfaction will be assessed separately with the visual analog scale. The value is between 0-10. A higher value indicates better satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Gonul Acar, PhD, Study Director — Marmara University; Hilal B Can, MSc, Principal Investigator — Marmara University
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No